CLINICAL TRIAL: NCT04251507
Title: The Use of Virtual Reality During Breast Localization Procedures
Brief Title: VR Ultrasound Guided Breast Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00092817
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2022-04

CONDITIONS: Breast Neoplasm Female
Keywords: Virtual Reality; Pain; Anxiety; Ultrasound Guided Needle Localization
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Goggles (Experimental): Patients randomized to the intervention group will undergo their procedure as standard of care but will wear the Oculus Go Goggles and experience a virtual reality simulation. The simulation is a non-interactive polar theme video.
  Interventions: Device: Oculus Go Virtual Reality Goggles
- Control (No Intervention): Patients randomized to the control group will undergo their procedure as standard of care without the use of virtual reality goggles.

INTERVENTIONS:
Device: Oculus Go Virtual Reality Goggles — Oculus Go is a standalone portable Virtual Reality device that enables the user to immerse in different virtual environments.Non pharmacological technique to reduce pain and anxiety during a procedure.
  Arms: Virtual Reality Goggles

SUMMARY:
To determine if a virtual reality simulation will reduce pain and anxiety in patients undergoing an ultrasound guided breast localization procedure (traditional wire, savi scout or a radiofrequency identification tag).

DETAILED DESCRIPTION:
Needle localizations for breast cancer surgery are required to identify cancerous tissue before surgery. Currently this procedure is done with or without a local anesthetic. Patients report anxiety regarding cancer and cancer-related procedures. Different types of needle localization may have different pain and anxiety based on their duration, complexity, and invasiveness. This research is designed to determine if VR simulated environment can reduce pain and anxiety.

Our aim is to study the efficacy of a virtual environment in reducing pain and procedural anxiety. It is intended for patients undergoing an ultrasound guided breast localization procedure that have had an abnormal breast biopsy. The overall aim is to discover an efficacious nonpharmacologic method to lower pain and anxiety during a standard of care procedure.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the patient
* Females ≥ 18 years of age
* Patient is schedule for preoperative ultrasound guided breast localization procedure

Exclusion Criteria:

* Patient is scheduled for or switched to a stereotactic localization procedure
* The patient has motion sickness
* The patient has severe cognitive disabilities or language barriers that inhibit study form completion in English
* Refusal of patient to sign consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Subjective Pain Assessment: Visual Analog Scale | Immediate post-procedure
  Pain Measured with the Visual Analog Scale. Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The individual will score their pain level by circling a number 0 - 10 at baseline, pre-operative, and post-operatively. The scale range includes 0-10 scales, with < 2 =well controlled, 2 - 5: partly controlled, > 5: uncontrolled.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI: Y-6 item) | Immediate post-procedure
  The State-Trait Anxiety Inventory uses a 4 point Likert scale to assess how much worry, tension or apprehension the subject experiences in his or her present circumstances (state anxiety) and how much anxiety represent a personality characteristic (trait anxiety). Items emphasize the frequency of particular symptoms (ranging from 1 = not at all to 4 = very much). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Patient Satisfaction | Immediate post-procedure
  Patients in both groups will be asked to rate their satisfaction with their procedures using a five point likert scale (ranging from 1 = definitely disagree to 5 = definitely agree).

OTHER OUTCOMES:
Heart Rate | Immediate post-procedure
  Empatica E4 watch is a wearable device that collects real-time physiological data. This wristband is equipped with photoplethysmogram sensors for computing Heart Rate (HR). Heart rate will be reported in beats per minute (bpm).
Temperature | Immediate post-procedure
  Empatica E4 watch is a wearable device that collects real-time physiological data. The photoplethysmogram sensor from the watch will measure temperature. Temperature will be reported in degrees Celsius.
Blood Volume Pulse Signal | Immediate post-procedure
  Empatica E4 watch is a wearable device that collects real-time physiological data. The photoplethysmogram sensor from the watch will measure variation of volume of arterial blood under the skin resulting from the heart cycle computing Blood Volume Pulse (BVP). Blood Volume Pulse will be measured in beats min-1.
Galvanic Skin Response | Immediate post-procedure
  The Empatica E4 watch is a wearable device that collects real-time physiological data. The photoplethysmogram skin electrodes from the watch will capture the Galvanic Skin Response (GSR), also named Electrodermal Activity (EDA) and Skin Conductance (SC) or the measure of the continuous variations in the electrical characteristics of the skin. GSR will be reported in units of micro-Siemens (μS).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Nisonson, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloomquist EV, Ajkay N, Patil S, Collett AE, Frazier TG, Barrio AV. A Randomized Prospective Comparison of Patient-Assessed Satisfaction and Clinical Outcomes with Radioactive Seed Localization versus Wire Localization. Breast J. 2016 Mar-Apr;22(2):151-7. doi: 10.1111/tbj.12564. Epub 2015 Dec 23. PMID 26696461
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Chirico A, Lucidi F, De Laurentiis M, Milanese C, Napoli A, Giordano A. Virtual Reality in Health System: Beyond Entertainment. A Mini-Review on the Efficacy of VR During Cancer Treatment. J Cell Physiol. 2016 Feb;231(2):275-87. doi: 10.1002/jcp.25117. PMID 26238976
- [Background] Costa WA, Monteiro MN, Queiroz JF, Goncalves AK. Pain and quality of life in breast cancer patients. Clinics (Sao Paulo). 2017 Dec;72(12):758-763. doi: 10.6061/clinics/2017(12)07. PMID 29319722
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Ratcliff CG, Prinsloo S, Chaoul A, Zepeda SG, Cannon R, Spelman A, Yang WT, Cohen L. A Randomized Controlled Trial of Brief Mindfulness Meditation for Women Undergoing Stereotactic Breast Biopsy. J Am Coll Radiol. 2019 May;16(5):691-699. doi: 10.1016/j.jacr.2018.09.009. Epub 2018 Oct 12. PMID 30322793
- [Background] Walker MR, Kallingal GJ, Musser JE, Folen R, Stetz MC, Clark JY. Treatment efficacy of virtual reality distraction in the reduction of pain and anxiety during cystoscopy. Mil Med. 2014 Aug;179(8):891-6. doi: 10.7205/MILMED-D-13-00343. PMID 25102532
- [Background] Wiederhold MD, Gao K, Wiederhold BK. Clinical use of virtual reality distraction system to reduce anxiety and pain in dental procedures. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):359-65. doi: 10.1089/cyber.2014.0203. PMID 24892198